CLINICAL TRIAL: NCT06090968
Title: Umbilical Cord Milking Versus Immediate Cord Clamping in Full Term Neonates (≥ 37 Weeks) Requiring Resuscitation - A RANDOMIZED CONTROL TRIAL
Brief Title: Umbilical Cord Milking Versus Immediate Cord Clamping in Full Term Neonates (≥ 37 Weeks) Requiring Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr. Sushma Nangia, Director Professor & Head, Department of Neonatology, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LHMC/IEC/071/UCM
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Perinatal Asphyxia
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord milking (Experimental): 20 cm of umbilical cord would be milked towards the infant with intact umbilical cord. The cord milking will be done four times. The entire procedure can be done in 15-20 seconds
  Interventions: Procedure: Umbilical cord milking
- Immediate cord clamping (Active Comparator): clamping the umbilical cord as soon as possible (average 30 seconds)
  Interventions: Procedure: Immediate cord clamping

INTERVENTIONS:
Procedure: Umbilical cord milking — 20 cm of umbilical cord would be milked towards the infant with intact umbilical cord. The cord milking will be done four times. The entire procedure can be done in 15-20 seconds
  Arms: Umbilical cord milking
Procedure: Immediate cord clamping — clamping the umbilical cord as soon as possible (average 30 seconds)
  Arms: Immediate cord clamping

SUMMARY:
The objective of the study is to compare the incidence of Hypoxic ischemic encephalopathy (all stages) among singleton term neonates (≥ 37 weeks) requiring resuscitation who will undergo Umbilical cord milking as compared to Immediate cord clamping.

DETAILED DESCRIPTION:
Enrolled participants will be randomly allocated to one of two study groups: 1) Umbilical cord clamping, 2) Immediate cord clamping

Umbilical cord clamping group: In the babies requiring resuscitation during vaginal delivery, the delivering obstetrician will place the infant on the mother's abdomen and about 20 cm of umbilical cord would be milked towards the infant with intact umbilical cord. The cord milking will be done four times by the obstetrical provider or by a second team member at the rate of 20 cm/2 sec. This procedure can be done in 15-20 seconds. Length of 20 cm can be estimated by the length of a sponge holding forceps which is approximately 25 cm. The umbilical cord will then clamped 2 -3 cm from the umbilical stump.

Immediate cord clamping: This will occur by clamping the umbilical cord as soon as possible (average 30 seconds).

Further resuscitation will be done in accordance with NRP 2015 guidelines. Stop watch will be used to calculate the duration after which the cord is clamped and cut, time to first breath, and time required to achieve HR > 100/min

ELIGIBILITY:
Inclusion Criteria:

Vaginally born, Singleton Term gestation (≥ 37 and & < 42 weeks), requiring resuscitation at birth

Exclusion Criteria:

* Major congenital anomaly (antenatally diagnosed or visible at birth)
* Rh negative pregnancy
* Hydrops
* Abruptio Placneta/ Placenta previa
* Fetus with absent and reversal of End Diastolic flow
* Cord avulsion
* Refusal of consent

Ages: 37 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypoxic Ischemic Encephalopathy | From date of birth until date of death from any cause whichever come first assessed till 1 week of life
  any stage as per Sarnat and Sarnat Staging

SECONDARY OUTCOMES:
Proportion requiring NICU admission | Till 1 week of life
  NICU admission due to any reason
Level of hypoxic ischemic encephalopathy ( mild, moderate or severe) | From date of birth until date of death from any cause whichever come first assessed till 1 week of life
  Level of hypoxic ischemic encephalopathy as per Sarnat and Sarnat Staging
Received blood products or saline bolus or inotropes to support blood pressure | From date of birth until date of death from any cause whichever come first assessed till 1 week of life
  Hypotension requiring blood products or saline bolus or inotropes
Length of hospital stay | From date of birth until date of death from any cause whichever come first assessed till 4 week of life
  Duration of stay in days
Mean Blood Pressure at 2,6,12,24,48,72 hrs | From date of birth until date of death from any cause whichever come first assessed till 72 hours of life
  Mean Blood Pressure as assessed by non-invasive oscillometric method
Hyperbilirubinemia requiring phototherapy | From date of birth until date of death from any cause whichever come first assessed till 4 week of life
  As per AAP charts
Proportion of neonates having APGAR score < 4 at 5 minutes of life | Till 5 minutes of life
  APGAR score (Min zero maximum Ten) assessed at 1,5 minutes (Low APGAR is bad prognosis and High APGAR is good prognosis)
Neonates requiring Initial steps of resuscitation, Bag and Mask Ventilation, Intubation, chest compression and administration of drugs during resuscitation. | Till 1 minutes of life
  As per NRP 2015 guidelines
Proportion of neonates developing polycythemia | Till first 72 hours
  Polycythemia is defined as venous hematocrit >65%
Proportion of mortality due to any cause | From date of birth until date of death from any cause whichever come first assessed till 4 week of life
  Including early and late neonatal deaths

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, DM (Neo), Study Chair — Lady Hardinge Medical College, New Delhi, India
Locations (1):
- Lady Hardinge Medical college, New Delhi, National Capital Territory of Delhi, India